CLINICAL TRIAL: NCT02626091
Title: Perfusion Evaluation by Real-time Fluorescence-based Enhanced Reality of Anastomosis
Acronym: PERFECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IHU Strasbourg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 15-005
Record Dates: First submitted 2015-12-03; First posted 2015-12-10 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Sigmoid Diverticulosis; Sigmoid Diverticulitis; Colorectal Malignancy
Keywords: Anastomotic perfusion; ICG Fluorescence; Enhanced reality; Left-sided colonic resection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Perfusion evaluation of anastomosis (Experimental): During left-sided colonic resections, anastomosis perfusion will be estimated by the visual appreciation of the surgeon and the ICG fluorescence-based enhanced reality. These two approaches will be compared.
  Interventions: Procedure: Left-sided colonic resection

INTERVENTIONS:
Procedure: Left-sided colonic resection — During interventions, anastomosis perfusion will be estimated (outcomes: visual appreciation of the surgeon, ICG fluorescence-based enhanced reality and series of peri-operative samplings) in order to validate the accuracy of ICG fluorescence-based enhanced reality technique.
  In any case, the resection will be performed according to the surgeon's appreciation.

SUMMARY:
The aim of this study is to evaluate the ability of a ICG-fluorescence guidance complemented with enhanced reality to correctly document intestinal pre-anastomotic perfusion and to validate the accuracy of this technique with metabolic intestinal cells changes.

DETAILED DESCRIPTION:
Accurate intraoperative evaluation of peri-anastomotic gastrointestinal tract perfusion is essential to reduce the risk of anastomotic complications such as leakage or strictures. Anastomotic leakage is the most dreadful complication of colorectal resections.

Intestinal microcirculation and viability is usually estimated from the color of the serosal surface, presence of peristalsis, pulsation and bleeding from the marginal arteries. This is subjective and based on the experience of the surgeon.

Fluorescence videography integrates a near-infrared endoscope able to detect the signal emitted by a fluorescent dye, Indocyanine Green (ICG), which is administered by intravenous injection. Fluorescence intensity is proportional to the amount of fluorescent dye diffused in the tissue and it consequently is a surrogate marker of tissue perfusion.

The hypothesis is that ICG-fluorescence guidance coupled with enhanced reality would allow a precise and rapid localization of the future anastomotic site in terms of optimal perfusion in laparoscopic colorectal resections.

In patients undergoing elective left-sided colonic resection by laparoscopic approach, resection site and anastomosis perfusion will be evaluated by :

* the visual appreciation of the surgeon
* the fluorescence-based enhanced reality, after injection of ICG and digital process.

A series of peri-operative samplings will also be carried out. In any case, the resection will be performed according to the surgeon's appreciation.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, from 18 years old
* Patient with sigmoid diverticulosis or diverticulitis
* Patient with colon malignancy
* Patient with rectum malignancy
* Patient with no contraindication to anesthesia and to colonic resection surgery
* Patient able to understand the study and to provide informed consent
* Patient affiliated to the French social security system

Exclusion Criteria:

* Patient undergoing emergency surgery
* Patient undergoing abdomino-perineal resection
* Patient undergoing colonic resection without anastomosis (Hartmann's colostomy)
* Patient with proven or unclear allergic reactions
* Pregnancy or breast-feeding
* Patient in exclusion period (determined by a previous study or in progress)
* Patient in custody
* Patient under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2018-09-14 (Actual); Study Completion 2018-09-14 (Actual)

PRIMARY OUTCOMES:
Correlation between the perfusion evaluated by the ICG fluorescence-based enhanced reality and the metabolic state of the intestine | During surgery
  The perfusion evaluated by the ICG fluorescence-based enhanced reality, obtained by the digital process of the fluorescence dynamic signal, will be correlated to the metabolic state of the intestine, assessed by the measure of biological markers on several points of the intestine.

SECONDARY OUTCOMES:
Correlation between the intraoperative intestinal perfusion and the rate of anastomosis leakage | During surgery
  The intraoperative intestinal perfusion on the anastomosis site, measured by fluorescence videography, will be correlated to the rate of anastomosis leakage.
Distance between the resection site based on the surgeon's appreciation and the resection site based on the digital analysis and the peri-operative samplings | During surgery
  The distance between the resection site based on the surgeon's clinic appreciation and the resection site based on the digital analysis and the level of capillary lactates and mitochondria respiratory rate on different sites will be measured.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Mutter, MD, PhD, Principal Investigator — Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil de Strasbourg; Michele Diana, MD, Study Director — IHU Strasbourg
Locations (1):
- Service de Chirurgie Digestive et Endocrinienne - Nouvel Hôpital Civil, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Diana M, Noll E, Diemunsch P, Dallemagne B, Benahmed MA, Agnus V, Soler L, Barry B, Namer IJ, Demartines N, Charles AL, Geny B, Marescaux J. Enhanced-reality video fluorescence: a real-time assessment of intestinal viability. Ann Surg. 2014 Apr;259(4):700-7. doi: 10.1097/SLA.0b013e31828d4ab3. PMID 23532109
- [Background] Diana M, Halvax P, Dallemagne B, Nagao Y, Diemunsch P, Charles AL, Agnus V, Soler L, Demartines N, Lindner V, Geny B, Marescaux J. Real-time navigation by fluorescence-based enhanced reality for precise estimation of future anastomotic site in digestive surgery. Surg Endosc. 2014 Nov;28(11):3108-18. doi: 10.1007/s00464-014-3592-9. Epub 2014 Jun 10. PMID 24912446
- [Background] Diana M, Dallemagne B, Chung H, Nagao Y, Halvax P, Agnus V, Soler L, Lindner V, Demartines N, Diemunsch P, Geny B, Swanstrom L, Marescaux J. Probe-based confocal laser endomicroscopy and fluorescence-based enhanced reality for real-time assessment of intestinal microcirculation in a porcine model of sigmoid ischemia. Surg Endosc. 2014 Nov;28(11):3224-33. doi: 10.1007/s00464-014-3595-6. Epub 2014 Jun 17. PMID 24935199
- [Background] Diana M, Agnus V, Halvax P, Liu YY, Dallemagne B, Schlagowski AI, Geny B, Diemunsch P, Lindner V, Marescaux J. Intraoperative fluorescence-based enhanced reality laparoscopic real-time imaging to assess bowel perfusion at the anastomotic site in an experimental model. Br J Surg. 2015 Jan;102(2):e169-76. doi: 10.1002/bjs.9725. PMID 25627131
- [Background] Boni L, David G, Mangano A, Dionigi G, Rausei S, Spampatti S, Cassinotti E, Fingerhut A. Clinical applications of indocyanine green (ICG) enhanced fluorescence in laparoscopic surgery. Surg Endosc. 2015 Jul;29(7):2046-55. doi: 10.1007/s00464-014-3895-x. Epub 2014 Oct 11. PMID 25303914
- [Derived] D'Urso A, Agnus V, Barberio M, Seeliger B, Marchegiani F, Charles AL, Geny B, Marescaux J, Mutter D, Diana M. Computer-assisted quantification and visualization of bowel perfusion using fluorescence-based enhanced reality in left-sided colonic resections. Surg Endosc. 2021 Aug;35(8):4321-4331. doi: 10.1007/s00464-020-07922-9. Epub 2020 Aug 27. PMID 32856153